CLINICAL TRIAL: NCT00138450
Title: Village Surveys of Morbidity Due to S. Haematobium for 1U01AI4547 Urinary Schistosomiasis-Determinants of Infection and Disease
Brief Title: Urinary Schistosomiasis Infection
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 01-588
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2007-03

CONDITIONS: Diseases of the Urinary System; Schistosomiasis Haematobia
Keywords: Schistosomiasis, S. haematobium, morbidity, Kenya
MeSH Terms: conditions — Urologic Diseases; Schistosomiasis haematobia; Schistosomiasis

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to determine what causes some people to become sick, and others not, when they are infected with the parasite Schistosoma haematobium, also known as Bilharzia. This is an infection of the urinary tract blood vessels and can cause serious disease. Approximately 4400 adults and children of any age will participate in this study. They must be residents of the Msambweni Area, Kwale District, Coast Province, Kenya, where infection with S. haematobium parasites are common. To find out if people are infected, they will first provide 1 or more urine samples for a microscope examination to detect if the S. haematobium parasites are present in the body. Volunteers then will be examined by ultrasound to see if they have kidney or bladder disease. (Ultrasound examination is the use of a non-painful machine that uses sound waves to examine the condition of the internal organs.) Treatment with the drug praziquantel will be offered if S. haematobium infection is found.

DETAILED DESCRIPTION:
The goal of this project is to focus both field and laboratory research on specific epidemiological, genetic and immunological features that underline the greatest susceptibility to S. haematobium infection and disease. This information, combined with epidemiological modeling of control strategies, will allow accelerated synthesis of the next generation of control programs. The studies in this initial Protocol A involve a large-scale survey of study villages to determine current population demography, general health, infection with S. haematobium, and, specifically, prevalence of parasite-related morbidity. Once evaluated, participants in Protocol A may be subsequently enrolled in Project Protocols B through F if they meet inclusion criteria. The size of the observational Protocol A study cohort (~4,400) is, in part, based on one of its secondary aims: i.e., the need to identify sufficient numbers of morbidity-concordant sibling pairs for genetic studies performed under Protocol D, and sufficient mother-infant pairs for Protocol F. Beyond initial screening, no further investigation occurs in Protocol A per se. Standard doses of praziquantel therapy will be given to treat S. haematobium infection diagnosed under Protocol A. Longitudinal follow-up of a subset of these treated individuals will be performed in Protocols B, C and E of the project. The study will enroll approximately 1100 adults and 1100 children from each of 2 types of rural S. haematobium-endemic village: a) those that have had prior participation in schistosomiasis control programs (1984-1993) and b) those that have not. The Msambweni area of Kwale District in southern Coast Province, Kenya will serve as the 'previously-treated' area. This area has participated in a long-term study of S. haematobium treatment since 1983. Three additional area villages (population ~4,000) that have not previously participated in treatment programs will be included as control 'previously-untreated' areas for comparison purposes to confirm the natural history of untreated infection. Like Msambweni area villages, the comparison villages (Mbuani, Mabakoni, and Gonjora) will be located in southern Kwale District, Coast Province, Kenya. In order to mirror the pre-control experience of the Msambweni villages, comparison villages will be selected primarily for their high S. haematobium prevalence (>40%) as determined in prior Ministry of Health sample surveys in schools. Secondary selection criteria will be village size (1200 to 2000 per village) and a rural, mostly agrarian environment. Residents will update their demography and kinship data, then receive physical examinations, urinalysis, ultrasound and parasitological examinations to determine infection and morbidity status. Because of its size, the population will be surveyed on a systematic, village-by village basis over the first 2 years of the project. These surveys will provide an effective cross-sectional evaluation of current levels of disease in treated and untreated communities at-large. Subjects with suspicion for severe renal dysfunction or bladder cancer (a known late complication of S. haematobium) will be referred to Msambweni or Mombasa Hospitals for further care. The primary study objective is to compare rates of moderate-to-severe urinary tract morbidity associated with S. haematobium infection for older children and adults residing in previously-treated and previously-untreated villages in the endemic southern Kwale District, Coast Province, Kenya. Secondary objectives are to: (1) compare rates of heavy S. haematobium infection for individuals residing in these previously-treated and -untreated villages; and (2) identify eligible subjects for participation in more detailed study of late S. haematobium-related disease, hereditary predisposition to morbidity, association of cytokine response to morbidity, and effects of in utero sensitization to S. haematobium on disease in later life (Protocols B-F of the project).

ELIGIBILITY:
Inclusion Criteria:

1. Kenyan residents, newborn to adult, either male or female.
2. Residence in areas of Kwale District endemic for Schistosoma haematobium

Exclusion Criteria:

Pregnancy (this is a partial exclusion). Pregnant women will participate in the parasitological screening phase of the study. However, because of pregnancy-related effects on the urinary system, their ultrasound examinations will be excluded from the analysis of hydronephrosis. Further, because of potential toxicity of praziquantel (Category B) and its alternative, metrifonate (an anticholinesterase), post-protocol anti-parasitic therapy will be delayed until the mother delivers and has stopped breastfeeding her infant.

Max Age: 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4400
Dates: Study Completion 2004-11

CONTACTS AND LOCATIONS:
Locations (1):
- KEMRI Centre for Geographic Medicine Research, Kilifi, Kenya